CLINICAL TRIAL: NCT02981056
Title: A Clinical Assessment of the Efficacy and Effects of Different Skincare Regimens on Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Collaborators: Beijing Children's Hospital (Other); Shanghai China-Norm Management Consulting co.,LTD (Unknown); Fudan University (Other); Shaanxi Bio-regenerative Biotechnology co.LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: JB-05-2012-31
Record Dates: First submitted 2016-11-30; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Baby Skin Development
Keywords: Skincare regimens; Skin moisturization; Skin barrier; Skin development
MeSH Terms: interventions — Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wash + Lotion regimen (Active Comparator): Johnson's Baby Top-To-Toe Wash (Ideally 7 times a week, at least 5 times a week) + Johnson's Baby Lotion (at least once a day).
  The products/treatment were used for a period of 3 months, and the products were placed on skin and with attention to applying the products on the arms, legs and torso.
  Interventions: Other: Johnson's Baby Top-To-Toe Wash; Other: Johnson's Baby Lotion
- Water + Lotion regimen (Active Comparator): Water (in lieu of bathing products) + Johnson's Baby Lotion (at least once a day).
  The products/treatment were used for a period of 3 months, and the products were placed on skin and with attention to applying the products on the arms, legs and torso.
  Interventions: Other: Johnson's Baby Lotion; Other: Water (in lieu of bathing products)
- Water only (Active Comparator): Water (in lieu of bathing products) only. The products/treatment were used for a period of 3 months, and the products were placed on skin and with attention to applying the products on the arms, legs and torso.
  Interventions: Other: Water (in lieu of bathing products)

INTERVENTIONS:
Other: Johnson's Baby Top-To-Toe Wash — During the study period, the different intervention products/regimens will be assigned to each group of subjects and replaced their daily wash and or body lotion products. Usage frequency: Ideally 7 times a week, at least 5 times a week, no more than once in the same day.
  Other Names: JB Wash
  Arms: Wash + Lotion regimen
Other: Johnson's Baby Lotion — During the study period, the different intervention products/regimens will be assigned to each group of subjects and replaced their daily wash and or body lotion products. Usage frequency: at least once a day, no more than twice in the same day.
  Other Names: JB Lotion
  Arms: Wash + Lotion regimen; Water + Lotion regimen
Other: Water (in lieu of bathing products) — During the study period, the different intervention products/regimens will be assigned to each group of subjects and replaced their daily wash and or body lotion products. Usage frequency: Ideally 7 times a week, at least 5 times a week, no more than once in the same day.
  Other Names: Water
  Arms: Water + Lotion regimen; Water only

SUMMARY:
The objective of the study is to investigate the effects of different skincare regimens on infants (0-6 months old at the start of the study), specifically focusing on moisturization effect. Outcome measures include moisturization, skin pH, skin barrier, physiological parameters, reactivity and skin microbiome.

DETAILED DESCRIPTION:
This is a single-center, single-blind, parallel study in healthy, full-term, male or female infants aged 0-6 months at the start of the study. The objective of the study is to investigate the effects of different skincare regimens on infants (0-6 months old at the start of the study), specifically focusing on moisturization effect. Outcome measures include moisturization, skin pH, skin barrier, physiological parameters, reactivity and skin microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Study Population: Healthy, full-term, male or female aged 0-6 months old at the start of the study. The newborn must not suffer from any pre-existing conditions (including skin conditions) that can adversely affect the outcome of the study.
2. The participating parent/legal guardian is the one who regularly cares for the newborn. This parent/legal guardian must be willing and able to follow all study directions, accept skin examination and commit to all follow-up visits for the duration of the study. The participating parent/legal guardian must agree to complete a daily diary, as well as questionnaires about use of the test product at each trial visit.

   1. For Cell No.1, the participating parent/legal guardian must be willing to bathe the newborn with the provided baby wash during every bath, at least 5 times a week throughout the remainder of the study. Test wash should be used no more than once in the same day.

      The participating parent/legal guardian must be willing to apply the provided test lotion at least once per day, in the morning. When bathing the newborn, the test lotion should be used after bathing. If the newborn is bathed in the afternoon or evening (at least 6 hours after the first lotion application), the test lotion is to be re-applied after bathing. Test lotion should be used no more than twice in the same day.
   2. For Cell No.2, the participating parent/legal guardian must be willing to bathe the newborn with water only during every bath, at least 5 times a week throughout the remainder of the study.

      The participating parent/legal guardian must be willing to apply the provided test lotion at least once per day, in the morning. When bathing the newborn, the test lotion should be used after bathing. If the newborn is bathed in the afternoon or evening (at least 6 hours after the first lotion application), the test lotion is to be re-applied after bathing. Test lotion should be used no more than twice in the same day.
   3. For Cell No.3, the participating parent/legal guardian must be willing to bathe the newborn with water only during every bath, at least 5 times a week throughout the remainder of the study but not more than once a day.

   The participating parent/legal guardian must be willing to not apply any body moisturizer to the newborn throughout the study.
3. The participating parent/legal guardian must be willing to read an IRB-approved informed consent agreement in Chinese, have all study related questions answered and to sign 2 copies of the agreement on behalf of his/her minor child (1 to retain and 1 for the study file).
4. Participating parent/legal guardian must be willing to complete a medical history and eligibility questionnaire related to his/her child, and to sign a photographic release, and a confidentiality agreement.
5. Participating parent/legal guardian must understand/agree that all of the following inclusion criteria must be met for 1 per household to be enrolled and participate in the study. One newborn in the household is eligible to participate in the study. Newborn is the only subject in the household who will participate in the study and routinely treated with the test materials alone.
6. Participating, adult parent/legal guardian of the subject must be 18 years of age or older and must be willing to present proof of guardianship (i.e., birth certificate, insurance card) at screening/baseline visit.
7. Participating parent/legal guardian must be willing to cooperate and participate by following study requirements for the duration of the study.
8. Participating parent/legal guardian must be willing to not bathe their newborn at least 12 hours prior to each clinic visit and to have the newborn wear loose-fitting clothing to each visit to accommodate procedures.
9. Participating parent/legal guardian must be willing for their newborn to have clean skin on baseline visit and all follow-up visits.
10. Parent/legal guardian must be willing to not apply any product to the newborn for 24 hours before visit until after the visit is completed.
11. Parent/legal guardian must be willing to replace the regular wash and lotion/moisturizer with the assigned products in this trial. Parent/legal guardian must continue to use newborn's regular brand of shampoo (but limit the use of shampoo on head/hair only), wipes/powder, and diaper rash ointment/cream as long as they have been using the product for at least 1 month prior to the start of the study.
12. Parent/legal guardian must agree not to use the provided test products on any other family member (other than the newborn participant) for the duration of the study.
13. Parent/legal guardian must be willing to use the product as a direct-to-skin with hand application. Parent/legal guardian must be willing to use the wash product without pouring it into the bath.
14. Parent/legal guardian must agree not to introduce any new fragrances on his/her person, or on his/her newborn (e.g. cleansers, lotions, perfumes, etc.), or in the household environment (e.g. room fresheners, cleansing agents, etc.) for the duration of the study.
15. Parent/legal guardian must agree not to expose his/her newborn participating in the study to excessive sun exposure. Parent/legal guardian must agree for the newborn to avoid extended sun exposure during the peak periods of 11 AM to 4 PM. If newborn is briefly exposed to the sun, parent/legal guardian will make every attempt to use protective clothing. No use of sunscreen is allowed throughout study participation.
16. Parent/legal guardian must agree not to permit their newborn from participating in another study for the duration of the study.
17. Parent/legal guardian must agree for the newborn to avoid the beach during the course of the study, and any activities at or in a swimming pool should be documented in the daily diary.
18. Evidence of a personally signed and dated Informed Consent document indicating that the Parent/legal guardian has been informed of all pertinent aspects of the trial.
19. Parent/legal guardian who is willing and able to comply with scheduled visits, study procedures, and other trial procedures.

Exclusion Criteria:

1. Any disease or condition of the skin (i.e. dermatitis, eczema, psoriasis, rosacea) that the Investigator deems inappropriate for participation.
2. Any newborn with clinically determined moderate to severe dryness (>2.0) or clinically determined erythema (>0.5), rash (>0.5), or an overall skin condition which, in the Investigator's judgment, makes the subject ineligible or places the subject at risk will not be enrolled in the study.
3. Any condition requiring use of a topical or oral OTC or prescription medication, which, in the investigator's judgment, makes the subject ineligible or places the subject at risk (e.g. antibiotics or any other medications that may cause gastrointestinal distress/diarrhea that will affect skin condition/cause irritation/rash of genital/buttocks area). Child vitamins are allowed and should be listed on the Medical Information sheet under the Concurrent Medications section.
4. Individuals currently involved in another clinical study of any type, or planning to participate in another clinical study of any type during this study.
5. Newborn participant who exhibits or is known to have atopic dermatitis, eczema, or other inflammatory disease, or mild to severe diaper rash or skin diseases/conditions that in the opinion of the investigator may affect the evaluation of study product or place the newborn at undue risk.
6. Newborn participant or parent/legal guardian who has experienced unusual hypersensitivity or allergic reactivity to fragrances and/or reaction/irritation to skin care toiletry products, or who has known allergies/sensitivities to ingredients in the provided test products.
7. Newborn participant or parent/legal guardian with a known condition of asthma or any related breathing problems and/or for whom there is a family history of asthma.
8. Newborn participant with chronic medical conditions or treatments that could interfere with the study or pose a risk to the newborn (including known immunodeficiency or lung related conditions).
9. Newborn participant with active localized or general infections including upper respiratory infections (ear, nose, throat, fever, cough, etc.).
10. Conditions that may interfere with the evaluation of the trial results, e.g., medical characteristics, diseases, or therapy that may interfere with the effect of the investigational product or with the evaluation of efficacy or safety variables. The conditions may also include concurrent use of another investigational product or prior use of an investigational product or approved medication or other drug within a defined period prior to trial enrollment.
11. Conditions for which subjects should be excluded for safety reasons, e.g., medical characteristics, disease, or therapy that may constitute contraindications or risks in connection with the use of the investigational product or the specified methods of evaluation.
12. Participation in other clinical trials within 30 days before the current trial begins and/or during trial participation
13. Other medical conditions that may increase the risk associated with trial participation or may interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial.
14. Parent/Legal guardian of the newborn is an employee of the investigator or study center or is a family member of the employees or the investigator.

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Skin surface moisture | 3 months
  Skin surface moisture content via capacitance measurements.

SECONDARY OUTCOMES:
Skin deep hydration | 3 months
  Skin deep Hydration and water content via measurement of dielectric constant of the skin to a depth of 500 microns.
Trans-epidermis water loss (TEWL) | 3 months
Ratio of TEWL/Skin surface moisture to reflect skin barrier function | 3 months
Skin pH value | 3 months
  Skin pH value measurement.
Skin roughness | 3 months
  Skin roughness estimated from digital images.
Dermatological assessments | 3 months
  Dermatological grading of overall skin condition, softness, dryness, redness (erythema), rash (irritation) and tactile roughness.
Parent/Caregiver assessments | 3 months
  Parent/Caregiver rating of overall skin condition, softness, dryness, redness (erythema), rash (irritation) and tactile roughness.
Skin microbiome | 3 months
  Skin microbiome analysis.
Skin bio-marker | 3 months
  Skin bio-marker analysis via tape stripping.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ma, PhD, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boireau-Adamezyk E, Baillet-Guffroy A, Stamatas GN. Age-dependent changes in stratum corneum barrier function. Skin Res Technol. 2014 Nov;20(4):409-15. doi: 10.1111/srt.12132. Epub 2014 Feb 12. PMID 24517174
- [Background] Nikolovski J, Stamatas GN, Kollias N, Wiegand BC. Barrier function and water-holding and transport properties of infant stratum corneum are different from adult and continue to develop through the first year of life. J Invest Dermatol. 2008 Jul;128(7):1728-36. doi: 10.1038/sj.jid.5701239. Epub 2008 Jan 17. PMID 18200056
- [Background] Stamatas GN, Nikolovski J, Mack MC, Kollias N. Infant skin physiology and development during the first years of life: a review of recent findings based on in vivo studies. Int J Cosmet Sci. 2011 Feb;33(1):17-24. doi: 10.1111/j.1468-2494.2010.00611.x. Epub 2010 Aug 30. PMID 20807257
- [Background] Walters RM, Khanna P, Chu M, Mack MC. Developmental Changes in Skin Barrier and Structure during the First 5 Years of Life. Skin Pharmacol Physiol. 2016;29(3):111-8. doi: 10.1159/000444805. Epub 2016 May 5. PMID 27161444
- [Background] Stamatas GN, Zerweck C, Grove G, Martin KM. Documentation of impaired epidermal barrier in mild and moderate diaper dermatitis in vivo using noninvasive methods. Pediatr Dermatol. 2011 Mar-Apr;28(2):99-107. doi: 10.1111/j.1525-1470.2011.01308.x. PMID 21504443
- [Background] Stamatas GN, Tierney NK. Diaper dermatitis: etiology, manifestations, prevention, and management. Pediatr Dermatol. 2014 Jan-Feb;31(1):1-7. doi: 10.1111/pde.12245. Epub 2013 Nov 14. PMID 24224482
- [Background] Blume-Peytavi U, Hauser M, Lunnemann L, Stamatas GN, Kottner J, Garcia Bartels N. Prevention of diaper dermatitis in infants--a literature review. Pediatr Dermatol. 2014 Jul-Aug;31(4):413-29. doi: 10.1111/pde.12348. Epub 2014 May 29. PMID 24890321
- [Background] Atherton D, Mills K. What can be done to keep babies' skin healthy? RCM Midwives. 2004 Jul;7(7):288-90. PMID 15314924
- [Background] Mack MC, Chu MR, Tierney NK, Ruvolo E Jr, Stamatas GN, Kollias N, Bhagat K, Ma L, Martin KM. Water-Holding and Transport Properties of Skin Stratum Corneum of Infants and Toddlers Are Different from Those of Adults: Studies in Three Geographical Regions and Four Ethnic Groups. Pediatr Dermatol. 2016 May;33(3):275-82. doi: 10.1111/pde.12798. Epub 2016 Feb 10. PMID 26860213
- [Background] Blume-Peytavi U, Lavender T, Jenerowicz D, Ryumina I, Stalder JF, Torrelo A, Cork MJ. Recommendations from a European Roundtable Meeting on Best Practice Healthy Infant Skin Care. Pediatr Dermatol. 2016 May;33(3):311-21. doi: 10.1111/pde.12819. Epub 2016 Feb 26. PMID 26919683
- [Background] Blume-Peytavi U, Hauser M, Stamatas GN, Pathirana D, Garcia Bartels N. Skin care practices for newborns and infants: review of the clinical evidence for best practices. Pediatr Dermatol. 2012 Jan-Feb;29(1):1-14. doi: 10.1111/j.1525-1470.2011.01594.x. Epub 2011 Oct 20. PMID 22011065
- [Background] Garcia Bartels N, Scheufele R, Prosch F, Schink T, Proquitte H, Wauer RR, Blume-Peytavi U. Effect of standardized skin care regimens on neonatal skin barrier function in different body areas. Pediatr Dermatol. 2010 Jan-Feb;27(1):1-8. doi: 10.1111/j.1525-1470.2009.01068.x. PMID 20199402
- [Background] Dizon MV, Galzote C, Estanislao R, Mathew N, Sarkar R. Tolerance of baby cleansers in infants: a randomized controlled trial. Indian Pediatr. 2010 Nov;47(11):959-63. doi: 10.1007/s13312-010-0161-8. Epub 2010 Mar 15. PMID 20453263
- [Background] Blume-Peytavi U, Cork MJ, Faergemann J, Szczapa J, Vanaclocha F, Gelmetti C. Bathing and cleansing in newborns from day 1 to first year of life: recommendations from a European round table meeting. J Eur Acad Dermatol Venereol. 2009 Jul;23(7):751-9. doi: 10.1111/j.1468-3083.2009.03140.x. PMID 19646134
- [Background] Gfatter R, Hackl P, Braun F. Effects of soap and detergents on skin surface pH, stratum corneum hydration and fat content in infants. Dermatology. 1997;195(3):258-62. doi: 10.1159/000245955. PMID 9407174
- [Background] Atrux-Tallau N, Huynh NT, Gardette L, Pailler-Mattei C, Zahouani H, Viviant E, Hirsch H, Marek H, Falson F, Pirot F. Effects of physical and chemical treatments upon biophysical properties and micro-relief of human skin. Arch Dermatol Res. 2008 Jun;300(5):243-51. doi: 10.1007/s00403-008-0849-y. Epub 2008 Apr 2. PMID 18386023
- [Background] Giusti F, Martella A, Bertoni L, Seidenari S. Skin barrier, hydration, and pH of the skin of infants under 2 years of age. Pediatr Dermatol. 2001 Mar-Apr;18(2):93-6. doi: 10.1046/j.1525-1470.2001.018002093.x. PMID 11358544
- [Background] Mayrovitz HN, Bernal M, Brlit F, Desfor R. Biophysical measures of skin tissue water: variations within and among anatomical sites and correlations between measures. Skin Res Technol. 2013 Feb;19(1):47-54. doi: 10.1111/srt.12000. Epub 2012 Oct 9. PMID 23046199
- [Background] Alanen E, Nuutinen J, Nicklen K, Lahtinen T, Monkkonen J. Measurement of hydration in the stratum corneum with the MoistureMeter and comparison with the Corneometer. Skin Res Technol. 2004 Feb;10(1):32-7. doi: 10.1111/j.1600-0846.2004.00050.x. PMID 14731246
- [Background] De Paepe K, Houben E, Adam R, Wiesemann F, Rogiers V. Validation of the VapoMeter, a closed unventilated chamber system to assess transepidermal water loss vs. the open chamber Tewameter. Skin Res Technol. 2005 Feb;11(1):61-9. doi: 10.1111/j.1600-0846.2005.00101.x. PMID 15691261
- [Background] Fluhr JW, Darlenski R, Lachmann N, Baudouin C, Msika P, De Belilovsky C, Hachem JP. Infant epidermal skin physiology: adaptation after birth. Br J Dermatol. 2012 Mar;166(3):483-90. doi: 10.1111/j.1365-2133.2011.10659.x. Epub 2012 Jan 19. PMID 21967466
- [Background] Saijo S, Tagami H. Dry skin of newborn infants: functional analysis of the stratum corneum. Pediatr Dermatol. 1991 Jun;8(2):155-9. doi: 10.1111/j.1525-1470.1991.tb00308.x. PMID 1923986
- [Background] Kvenshagen B, Jacobsen M, Halvorsen R. Atopic dermatitis in premature and term children. Arch Dis Child. 2009 Mar;94(3):202-5. doi: 10.1136/adc.2008.142869. Epub 2008 Oct 1. PMID 18829619